CLINICAL TRIAL: NCT05274659
Title: A Randomized, Single-blinded, Placebo Controlled, Single Ascending Dose Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of KJ103 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety and Tolerability of KJ103 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Bao Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHBJ-2021-001
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- KJ103 dose group 1 (Active Comparator): KJ103 single dose
  Interventions: Drug: KJ103
- KJ103 dose group 2 (Active Comparator): KJ103 single dose
  Interventions: Drug: KJ103
- KJ103 dose group 3 (Active Comparator): KJ103 single dose
  Interventions: Drug: KJ103
- KJ103 dose group 4 (Active Comparator): KJ103 single dose
  Interventions: Drug: KJ103
- KJ103 dose group 5 (Active Comparator): KJ103 single dose
  Interventions: Drug: KJ103
- Matching placebo for each dose group (Placebo Comparator): placebo, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KJ103 — Recombinant Immunoglobulin G Cleaving Enzyme
  Other Names: no other invention names
  Arms: KJ103 dose group 1; KJ103 dose group 2; KJ103 dose group 3; KJ103 dose group 4; KJ103 dose group 5
Drug: Placebo — Placebo
  Other Names: no other invention names
  Arms: Matching placebo for each dose group

SUMMARY:
This is a randomized, single-blinded, placebo controlled, single ascending dose phase I study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) and immunogenicity of KJ103 in healthy subjects.

DETAILED DESCRIPTION:
This single ascending dose (SAD), randomized, single-blinded, placebo controlled study is the first study and it is designed to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of KJ103 in healthy subjects after a single intravenous dose. It will include up to 34 healthy subjects in up to five dose groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 55 years, inclusive.
2. Male body weight ≥50kg, female body weight ≥45kg, body mass index (BMI) within 18 kg/m2to 35 kg/m2, inclusively.
3. Immunoglobulin (IgG) levels at screening is within the normal range.
4. Considered "healthy" by the investigator. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, as well as a complete physical examination including vital signs, 12-lead ECG, hematology, biochemistry, and urinalysis.

Exclusion Criteria:

1. History of or diagnosis at screening of any clinically significant immunodeficiency including but not limited to immunoglobulin A deficiency.
2. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease.
3. Any clinically significant illness in the 28 days prior to the first study drug administration.
4. Any history of tuberculosis.
5. Positive screening results to HIV Ag/Ab combo, syphilus, hepatitis A, hepatitis B surface antigen or hepatitis C virus tests.
6. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration.
7. Current use of tobacco or nicotine-containing products exceeding 10 cigarettes per day or equivalent.
8. Received an investigational drug (or was using an investigational device at the time) within 30 days prior to screening, or at least 5 times the respective elimination half-life (if known), whichever is longer.
9. Female who is lactating.
10. Female who is pregnant according to the pregnancy test at screening or prior to the first study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
AE | Day 1 through Day 14
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational drug

SECONDARY OUTCOMES:
Cmax | Up to 144 hours postdose
  The maximum measured concentration of the analysis in serum
Tmax | Up to 144 hours postdose
  Time To Reach The Maximal serum Concentration
t½ | Up to 144 hours postdose
  Terminal Elimination Half-Life
AUC0-inf | Up to 144 hours postdose
  Area Under the Serum Concentration Versus Time Curve From Zero to Infinity
IgG level | Day 1 through Day 63
  Concentration of Immunoglobulin G in serum

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hamilton, Principal Investigator — New Zealand Clinical Research
Locations (1):
- New Zealand Clinical Research, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No